CLINICAL TRIAL: NCT01312415
Title: A Comparison of the Analgesic Efficacy of Local Anaesthetic Wound Infiltration Versus Intrathecal Morphine for Total Knee Replacement
Brief Title: The Analgesic Efficacy of Local Anaesthetic Wound Infiltration Versus Intrathecal Morphine for Total Knee Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cork University Hospital (Other)
Responsible Party: Denise McCarthy, Anaesthesia Specialist Registrar, Cork University Hospital, Cork, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKR-SMOH
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Total Knee Replacement
Keywords: total knee arthroplasty; total knee replacement; local infiltration analgesia; intra-articular local anaesthesia; patients undergoing total knee arthroplasty (total knee replacement)
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- levobupivacaine infiltration (Experimental): Patients will receive spinal anaesthesia with intrathecal bupivacaine (17.5 or 15 mg) without morphine, and will receive peri- and intraarticular surgical site infiltration before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight (maximum 200mg levobupivacaine) plus 0.5mg epinephrine made up to 100ml with saline. An intra-articular catheter will be placed by the surgeon before closure under the sterile surgical conditions and this will be left in situ in the wound. The patient will receive one further injection of 15ml of levobupivacaine 0.5% at 8am the following morning.
  Interventions: Drug: Levobupivacaine
- Control (Other): Patients will receive spinal anaesthesia with intrathecal bupivacaine 0.5% (17.5 mg if greater than 70 kg and 15 mg if less than 70 kg) and preservative-free morphine (0.3 mg).
  Interventions: Drug: Intrathecal morphine

INTERVENTIONS:
Drug: Levobupivacaine — Patients will receive peri- and intraarticular surgical site infiltration to the knee during surgery and before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight (maximum 200mg levobupivacaine will be used if the patient's weight exceeds 100kg) plus 0.5mg epinephrine made up to 100ml with saline. An intra-articular catheter will be placed by the surgeon before closure under the sterile surgical conditions and this will be left in situ in the wound. The patient will receive one further injection of 15ml of levobupivacaine 0.5% solution at 8am on the morning of the first postoperative day after which the catheter will be removed.
  Arms: levobupivacaine infiltration
Drug: Intrathecal morphine — Patients will receive spinal anaesthesia with intrathecal bupivacaine 0.5% (17.5 mg if greater than 70 kg and 15 mg if less than 70 kg) and preservative-free morphine (0.3 mg).
  Arms: Control

SUMMARY:
Total knee replacement (TKR) is associated postoperatively with considerable pain and analgesic requirement. Total knee replacement is routinely performed under spinal anaesthesia with intrathecal bupivacaine plus preservative free morphine. We hypothesize that infiltration of the surgical site with peri- and intraarticular levobupivacaine local anaesthetic would be an efficacious pain management technique and would not be inferior to intrathecal morphine for postoperative pain management.

We further hypothesize that the use of this surgical site infiltration technique would decrease post-operative systemic opioid requirements as well as the side effects associated with intrathecal and systemic opioids.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral total knee replacement
* Consent to spinal anaesthesia
* ASA Grade I to III

Exclusion Criteria:

* Patient refusal
* Mini-Mental Score < 25 (see appendix 3)
* Allergy to bupivacaine, morphine, paracetamol, diclofenac
* Skin lesions/infection at site of injection
* Uncorrected renal dysfunction
* Coagulation disorders
* chronic pain condition other than knee pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Quality of analgesia in the postoperative period as assessed by visual analogue score (VAS) for pain at rest and on movement | 24 hours postoperatively

SECONDARY OUTCOMES:
Opioid consumption in total in the first 48 hours postoperatively | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Denise M McCarthy, MB FCARSCI, Principal Investigator — Cork University Hospital
Locations (1):
- St Mary Orthopedic Hospital, Cork, Ireland

REFERENCES:
- [Derived] McCarthy D, McNamara J, Galbraith J, Loughnane F, Shorten G, Iohom G. A comparison of the analgesic efficacy of local infiltration analgesia vs. intrathecal morphine after total knee replacement: A randomised controlled trial. Eur J Anaesthesiol. 2019 Apr;36(4):264-271. doi: 10.1097/EJA.0000000000000943. PMID 30640244